CLINICAL TRIAL: NCT03993483
Title: Variability in Resistance Training-induced Hypertrophy and Strength Are Independent of Load and Limb Location in Healthy Young Men
Brief Title: Upper Versus Lower Limb Responses to Higher Versus Lower Load Resistance Training in Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Tier 1 Canada Research Chair and Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HIREB 4774
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Muscle Hypertrophy; Muscle Strength

STUDY DESIGN:
Intervention Model Description: One arm and one leg of each participant were randomized to lift with heavier loads while the other arm and leg of each participant were randomized to lift with lighter loads for 10 weeks.
Who Masked: Outcomes Assessor
Masking Description: The histochemistry and ultrasonography were analyzed by blinded study investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher Load (Experimental): One arm and one leg were randomized (based on limb dominance) to perform unilateral biceps curls (arm) and knee extensions (leg) with relatively higher loads (80 % of their one-repetition maximum).
  Interventions: Behavioral: Unilateral resistance exercise
- Lower Load (Experimental): The other arm and leg were randomized (based on limb dominance) to perform unilateral biceps curls (arm) and knee extensions (leg) with relatively higher loads (80 % of their one-repetition maximum).
  Interventions: Behavioral: Unilateral resistance exercise

INTERVENTIONS:
Behavioral: Unilateral resistance exercise — The participants performed three sets of their unilateral resistance exercise (biceps curls and knee extensions) three times per week for 10 weeks.

SUMMARY:
Recent research suggests that performing resistance exercise training with relatively light loads is equally as effective at increasing muscle mass and muscle strength as performing resistance exercise training with relatively heavy loads. Whether or not performing resistance exercise with relatively heavy loads or light loads is equally as effective between the upper- and lower-body within the same individual has never been investigated. Given the substantial individual variance in resistance exercise training-induced changes in muscle mass and strength, this study is designed to quantify the relative influence that extrinsic training variables (e.g., load), as opposed to intrinsic muscle-based predisposition, has on resistance training-induced changes in muscle mass and muscle strength.

DETAILED DESCRIPTION:
Each participant will come to the Exercise Metabolism Research Laboratory gym three times per week for 10 weeks to perform lower- and upper-body resistance exercise training with both relatively heavy- (~80% one repetition maximum [1RM]) and light- (~40 %1RM) loads. One arm and one leg will be randomized to lift with relatively heavy loads such that the other arm and leg will be randomized to lift with relatively light loads. Each workout will be supervised by a study investigator.

The time commitment of this study is 12 weeks (including pre- and post-study testing). Each workout to take 30 minutes and, with testing days included, the investigators foresee a total time commitment of 41 hours, or just under three and half hours per week.

The pre- and post-study measurements include muscle biopsies, dual x-ray absorptiometry scans, ultrasonography scans, 1RM assessment, and maximum voluntary contraction assessment. The muscle biopsies will be taken from each of the participant's vastus lateralis to assess muscle fibre cross sectional area in both legs during the beginning (four biopsies) and end (four biopsies) of the intervention. The dual x-ray absorptiometry scans are used to assess body composition and will be done pre- and post-intervention. The ultrasonography scans will be used to assess biceps brachii and vastus laterals thickness and cross sectional area. The ultrasound scans will be assessed during the beginning (four scans) and end (four scans) of the intervention. The 1RM assessment will include 1RM testing on a knee extension machine and biceps curl machine and will be done at the beginning and end of the intervention. The maximum voluntary contraction assessment will be performed on a System 3 Biodex Dynamometer (Shirley, NY, USA), which is an immovable machine that the participants contract against to measure their peak force. The maximum voluntary contractions will be recorded three times: twice at the beginning of the intervention and once at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-30 years (inclusive)
* Be able to maintain a habitual diet and perform resistance exercise three times per week throughout the trial
* Be in general good health (assessed by Get Active Questionnaire)
* Understand the study procedures and sign this form providing informed consent to participate in the study.

Exclusion Criteria:

* Use of tobacco or related products
* A history of neuromuscular problems or muscle and/or bone wasting diseases
* Any acute or chronic illness; cardiac, pulmonary, liver, or kidney abnormalities; insulin- or non-insulin-dependent diabetes or other metabolic disorders (all ascertained through medical questionnaires)
* Use of medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatory drugs (prescription use or daily use of over the counter medication), or prescription strength acne medications)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Change in fat-free mass | up to 12 weeks
  Measured by dual x-ray absorptiometry pre- and post-training
Change in vastus lateralis thickness | up to 12 weeks
  Measured by ultrasonography pre- and post-training
Change in vastus lateralis cross sectional area | up to 12 weeks
  Measured by ultrasonography pre- and post-training
Change in biceps brachii thickness | up to 12 weeks
  Measured by ultrasonography pre- and post-training
Change in biceps brachii cross sectional area | up to 12 weeks
  Measured by ultrasonography pre- and post-training
Change in muscle fibre cross sectional area | up to 12 weeks
  Measured by muscle biopsies from the vastus lateralis pre- and post-training

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers